CLINICAL TRIAL: NCT07365215
Title: Pediatric Delirium in Swedish PICUs: Incidence, Risk Factors, and Validation of the Swedish Cornell Assessment of Pediatric Delirium (CAPD) Instrument.
Brief Title: Pediatric Delirium in Swedish Paediatric Intensive Care Units
Acronym: PADI
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Vastra Gotaland Region (Other Government); Region Skane (Other); Uppsala University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-01737-01
Record Dates: First submitted 2025-11-14; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Delirium; Pediatric Intensive Care; Risk Factors
Keywords: Pediatric Delirium; Delirium Assessment; PICU; Pediatric intensive care unit; Incidence; Risk Factors; CAPD; Cornell Assessment of Pediatric Delirium; Critical Care; Children; Sweden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to determine the incidence of delirium among children in a pediatric intensive care unit (PICU) and to identify associated risk factors.

Research Questions:

What is the incidence of delirium among children in a pediatric intensive care unit? What are the identifiable risk factors that predispose children in a pediatric intensive care unit to developing delirium?

DETAILED DESCRIPTION:
Study Background and Rationale Delirium, an acute neurocognitive syndrome, is characterized by a sudden onset of fluctuating mental states, reflecting a deterioration in brain function. Its clinical manifestations include impaired attention span, sleep disturbances, acute confusion, impaired concentration, decreased level of consciousness and responsiveness, increased irritability, apathy, or agitation. The duration of delirium can vary from short periods to several days and may fluctuate throughout hospitalization. The presence of delirium can significantly contribute to an increased length of hospital stay and can exacerbate suffering for both the pediatric patient and their family. In Swedish pediatric intensive care units (PICUs), a systematic assessment of delirium using a standardized, validated assessment instrument has historically been absent. This gap in practice hinders the early identification of affected children, which is crucial for improving care and mitigating adverse outcomes. Recognizing this need, an assessment instrument, the Cornell Assessment of Pediatric Delirium (CAPD), has been rigorously translated and culturally adapted from English to Swedish. This study is designed to implement this newly translated instrument to establish the incidence of delirium in children within Swedish PICUs. Furthermore, a critical objective is to identify associated risk factors, which will inform the development and implementation of targeted care strategies aimed at reducing the risk and burden of delirium. The proactive assessment and management of delirium are well-established standard practices in adult intensive care settings, underscoring the imperative for similar advancements in pediatric critical care.

Study Objectives and Research Questions Aim: This observational study aims to determine the incidence of delirium among children in a pediatric intensive care unit (PICU) and to identify associated risk factors.

Research Questions

* What is the incidence of delirium among children in pediatric intensive care units?
* What are the identifiable risk factors that predispose children in a pediatric intensive care unit to developing delirium?

Study Design and Setting This is a prospective, longitudinal multicenter observational study conducted across multiple pediatric intensive care units in Sweden. The study design is optimized for capturing real-world data on delirium incidence and associated factors in a diverse PICU population.

Participant Eligibility Participant eligibility criteria are comprehensively detailed in a separate protocol section. Briefly, the study will include children admitted to participating PICUs with an expected duration of care exceeding one over night stay. The primary consideration for inclusion is the ability for children (with assent as appropriate) and/or their parents/legal guardians to be informed about the study's purpose and provide consent. A deferred consent procedure will be utilized in emergency situations preventing immediate consent, wherein provisional inclusion occurs, followed by formal consent/assent at the earliest calm moment. In cases of consent withdrawal, all previously collected data for that participant will be immediately destroyed. Given the observational nature of the study, without any direct intervention, the risk of privacy violation under the deferred consent procedure is considered minimal.

Study Procedures and Data Collection Prior to the commencement of data collection, comprehensive education regarding pediatric delirium and the standardized administration of the CAPD instrument will be delivered to all nursing staff in participating PICUs. This initial training will ensure consistent application of the assessment tool across all sites. Continuous training modules will also be available for newly hired staff and accessible on demand, through both in-person sessions and remote online platforms, to maintain proficiency and adherence to protocol.

Delirium Assessment Following ethical approval, CAPD assessments will be systematically performed once per nursing shift for all eligible children admitted to the unit. This assessment will continue for each participant for a period of up to 24 months.

Clinical Data Elements

In addition to the CAPD assessment for delirium incidence, a comprehensive set of clinical data will be collected through direct inquiry with treating staff and through detailed electronic health record (EHR) review. Data elements considered relevant for identifying risk factors for delirium, characterizing delirium subtypes, and calculating delirium duration include, but are not limited to:

* Demographics: Age (at admission), gender.
* Medical History: Documented pre-existing conditions (e.g., neurological disorders, developmental delays).
* Clinical Course Data: Laboratory analyses (e.g., inflammatory markers, electrolyte levels, drug levels). Diagnostic findings (e.g., neurological diagnoses, infection status). Functional assessments (e.g., baseline functional status, mobility). Imaging results (e.g., cranial CT/MRI findings). Physiological Parameters: Continuously recorded vital signs (e.g., blood pressure, heart rate, respiratory rate, oxygen saturation), urine output, pain scores. Complications: Documented occurrences of renal failure, thrombotic events, episodes of decreased level of consciousness. Treatments: Initiation and duration of therapies such as dialysis, mechanical ventilation, specific medications (e.g., sedatives, analgesics, corticosteroids, vasopressors, anti-infectives). Nursing Interventions: Use of physical restraints, documented parental presence at the bedside, environmental modifications.

Data Management System Data will be collected by PICU nurses during the delirium assessment and subsequently managed by a designated research contact (1-2 persons) at each unit. All collected data will be entered into a secure, validated electronic Case Report Form (eCRF) database. Initial data will be captured via CAPD scores and select clinical variables. Subsequent retrospective EHR review will complement this initial dataset, with additional relevant clinical and historical data collected and entered into the same eCRF database.

Data Dictionary A comprehensive data dictionary will be maintained, providing detailed descriptions of each variable collected within the eCRF. This includes variable names, definitions, data types, allowable ranges, coding information (e.g., ICD-10 codes, MedDRA terms if applicable), and normal physiological ranges where relevant. The source of each variable (e.g., CAPD score, EHR abstraction) will also be documented.

Standard Operating Procedures (SOPs)

Detailed SOPs will govern all aspects of the study operations and analysis activities, including:

* Patient recruitment and screening.
* Informed consent/assent procedures, including deferred consent.
* Standardized CAPD assessment administration.
* Clinical data collection and EHR abstraction.
* Data entry into the eCRF.
* Data management, including data cleaning and validation.
* Handling and reporting of adverse events (if any related to study procedures).
* Change management for protocol amendments.

Study Staff Roles Each pediatric intensive care unit will designate 1-2 nurses primarily responsible for patient inclusion, informed consent processes, and consistent CAPD assessments. Additionally, a research assistant or nurse will be allocated to assist with meticulous EHR review and data entry to ensure accuracy and completeness. Permissions for EHR review will be formally sought from each participating hospital in accordance with local regulations and ethical guidelines.

Quality Assurance and Data Integrity Data entered into the eCRF system will undergo manual validation by personnel independent of the primary data collection team. A minimum of 10% of the entered records will be thoroughly reviewed. This manual review, will include assessment of data ranges, formats, and consistency across related data fields to minimize entry errors.

Source Data Verification (SDV) A proportion of the eCRF data, particularly critical variables related to delirium incidence and key risk factors, will undergo source data verification by comparing it against original medical records (EHRs). This will assess the accuracy and representativeness of the registry data.

Site Monitoring and Auditing Regular monitoring visits (remote or on-site, as determined by the study's scope and resources) will be conducted to ensure protocol adherence, proper CAPD administration, and data quality. Independent auditing may be performed to ensure compliance with regulatory and ethical standards.

Statistical Analysis Plan The sample size assessment will be performed to ensure adequate statistical power for the primary objectives, particularly for estimating the incidence of delirium with a specified precision and for identifying significant risk factors through multivariable logistic regression.

A plan will address missing data. Strategies for handling missing variables will include: Documentation of reasons for missingness. Assessment of patterns of missing data (e.g., Missing Completely at Random, Missing at Random, Missing Not at Random). Implementation of appropriate imputation techniques (e.g., multiple imputation) if deemed necessary and justifiable, following sensitivity analyses to assess the impact of missing data.Data will be analyzed using standard statistical software.

Descriptive Statistics Baseline characteristics of the study population will be summarized using descriptive statistics (e.g., means with standard deviations or medians with interquartile ranges for continuous variables; frequencies and proportions for categorical variables). The incidence of delirium will be presented as a proportion of children experiencing at least one episode of delirium during their PICU stay, along with its 95% confidence interval. The cumulative duration of delirium will be described using measures such as mean, median, and range of days. Delirium subtypes (hypoactive, hyperactive, mixed) will be reported using frequencies and proportions.

Inferential Statistics To identify risk factors, multivariable logistic regression models will be constructed. To explore associations with delirium duration, linear regression or other generalized linear models will be considered. Associations between risk factors and delirium subtypes may be analyzed using multinomial logistic regression or chi-square tests. Potential covariates, including demographic, clinical, and treatment-related factors identified during data collection, will be considered for inclusion in the models. Model selection will be based on established statistical criteria. Subgroup analyses may be performed if indicated by the data. All statistical tests will be two-sided, with a significance level set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

• Expected time of care at the pediatric intensive care unit for at least one overnight stay

Exclusion Criteria:

• Care at the very end of life

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children admitted to a pediatric intensive care unit with an expected time of care for at least one over night stay
Sampling Method: Non-Probability Sample
Enrollment: 676 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Delirium | Up to 24 months from PICU admission.
  This measure reports the proportion of participants who experience at least one episode of delirium during their pediatric intensive care unit (PICU) stay. Delirium is defined as an acute change in mental status characterized by impaired attention, disorganized thinking, or altered consciousness. Delirium will be determined by daily, once-per-shift assessments using the Cornell Assessment of Pediatric Delirium (CAPD) instrument, a validated bedside screening tool administered by trained nurses. A CAPD score of 9 or higher (on a scale of 0-32, with higher scores indicating greater delirium severity) will be considered indicative of delirium.

SECONDARY OUTCOMES:
Identification of Risk Factors for Delirium | Up to 24 months from PICU admission.
  This outcome will identify specific demographic, clinical, physiological, and treatment-related characteristics that increase the likelihood of developing delirium. Variables to be assessed for their association with delirium include, but are not limited to, patient age, gender, underlying medical conditions, physiological parameters (e.g., vital signs, lab values), administered medications (e.g., sedatives, opioids), and nursing interventions (e.g., use of restraints, parental presence). Associations will be determined through multivariable logistic regression analyses, identifying statistically significant predictors of delirium occurrence.
Cumulative Duration of Delirium | Up to 24 months from PICU admission.
  This outcome reports the total number of days (or shifts) during which a participant meets the criteria for delirium (CAPD score of 9 or higher) during their PICU stay. This measure quantifies the cumulative burden of delirium for each child, calculated by summing all days/shifts where a CAPD score of 9 or higher was recorded.
Delirium Subtype Characterization (Hypoactive, Hyperactive, Mixed) | Up to 24 months from PICU admission.
  This outcome will characterize delirium episodes based on their clinical presentation as hypoactive, hyperactive, or mixed subtypes. Hypoactive delirium is characterized by lethargy, reduced motor activity, and apathy, while hyperactive delirium presents with agitation, restlessness, and hyper-alertness. Mixed delirium includes features of both. Subtype classification will be based on specific criteria derived from nursing observations recorded alongside the CAPD assessments, potentially utilizing relevant CAPD item scores related to psychomotor activity.

CONTACTS AND LOCATIONS:
Overall Officials: Ylva Therström Blomqvist, Assoc Prof, Study Director — Uppsala University, Department of Women's and Children's Health
Locations (3):
- Sweden (3):
  - BIVA Göteborg, Gothenburg
  - BIVA Lund, Lund
  - BIVA Uppsala, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in publications from this study will be made available. This will include baseline characteristics, clinical course variables (such as physiological parameters, laboratory analyses, diagnostic findings, and complications), treatment exposures (e.g., medications, mechanical ventilation, nursing interventions), and delirium outcome data (incidence, cumulative duration, and subtype characterization based on CAPD assessments). All data will be fully anonymized at the individual level so that no participant can be identified.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 12 months after publication of the primary results and will remain available upon reasonable request for at least 5 years thereafter.
Access Criteria: Access to the de-identified dataset will be granted to qualified researchers upon reasonable request. Requests must include a brief description of the research question, analysis plan, and intended use of the data. All requests will be reviewed by the PADI steering committee. Data will be shared only for scientifically sound projects and for purposes consistent with the original study objectives and ethical approvals. Data will be shared through secure data transfer following approval of a data sharing agreement. No direct identifiers or site-specific identifiers will be included in the shared dataset.

REFERENCES:
- [Background] Thibault C, Pont-Thibodeau GD, MacDonald S, Jutras C, Metras ME, Harrington K, Toledano B, Roumeliotis N, Farrell C, Lacroix J, Ducharme-Crevier L. Two months outcomes following delirium in the pediatric intensive care unit. Eur J Pediatr. 2024 Jun;183(6):2693-2702. doi: 10.1007/s00431-024-05491-w. Epub 2024 Mar 23. PMID 38520519
- [Background] Dervan LA, Killien EY, Smith MB, Watson RS. Health-Related Quality of Life Following Delirium in the PICU. Pediatr Crit Care Med. 2022 Feb 1;23(2):118-128. doi: 10.1097/PCC.0000000000002813. PMID 34534165
- [Background] Ge XH, Wei WR, Feng TN, Xu LL, Hu YQ, Yuan CR. Analysis of risk factor for pediatric intensive care unit delirium in children: a case-control study. Am J Transl Res. 2021 Aug 15;13(8):9143-9151. eCollection 2021. PMID 34540029
- [Background] Semple D, Howlett MM, Strawbridge JD, Breatnach CV, Hayden JC. A Systematic Review and Pooled Prevalence of Delirium in Critically Ill Children. Crit Care Med. 2022 Feb 1;50(2):317-328. doi: 10.1097/CCM.0000000000005260. PMID 34387241
- [Background] Harris J, Ramelet AS, van Dijk M, Pokorna P, Wielenga J, Tume L, Tibboel D, Ista E. Clinical recommendations for pain, sedation, withdrawal and delirium assessment in critically ill infants and children: an ESPNIC position statement for healthcare professionals. Intensive Care Med. 2016 Jun;42(6):972-86. doi: 10.1007/s00134-016-4344-1. Epub 2016 Apr 15. PMID 27084344
- [Background] Pilato TC, Mauer EA, Gerber LM, Traube C. Pediatric Delirium and All-Cause PICU Readmissions Within 1 Year. Pediatr Crit Care Med. 2022 Oct 1;23(10):766-773. doi: 10.1097/PCC.0000000000003037. Epub 2022 Jul 27. PMID 35894610
- [Background] Siegel EJ, Traube C. Pediatric delirium: epidemiology and outcomes. Curr Opin Pediatr. 2020 Dec;32(6):743-749. doi: 10.1097/MOP.0000000000000960. PMID 33105274
- [Background] Smith HAB, Besunder JB, Betters KA, Johnson PN, Srinivasan V, Stormorken A, Farrington E, Golianu B, Godshall AJ, Acinelli L, Almgren C, Bailey CH, Boyd JM, Cisco MJ, Damian M, deAlmeida ML, Fehr J, Fenton KE, Gilliland F, Grant MJC, Howell J, Ruggles CA, Simone S, Su F, Sullivan JE, Tegtmeyer K, Traube C, Williams S, Berkenbosch JW. 2022 Society of Critical Care Medicine Clinical Practice Guidelines on Prevention and Management of Pain, Agitation, Neuromuscular Blockade, and Delirium in Critically Ill Pediatric Patients With Consideration of the ICU Environment and Early Mobility. Pediatr Crit Care Med. 2022 Feb 1;23(2):e74-e110. doi: 10.1097/PCC.0000000000002873. PMID 35119438
- [Background] Traube C, Silver G, Kearney J, Patel A, Atkinson TM, Yoon MJ, Halpert S, Augenstein J, Sickles LE, Li C, Greenwald B. Cornell Assessment of Pediatric Delirium: a valid, rapid, observational tool for screening delirium in the PICU*. Crit Care Med. 2014 Mar;42(3):656-63. doi: 10.1097/CCM.0b013e3182a66b76. PMID 24145848
- [Background] Xu TT, Zhang YC, Ye XF, Fu CH, Li Y, Ju MJ, Liu J, Yang XY, Zhang WY. Risk factors of delirium in a paediatric intensive care unit: A prospective case series study. Nurs Crit Care. 2023 Sep;28(5):645-652. doi: 10.1111/nicc.12920. Epub 2023 Apr 26. PMID 37186353
- [Background] Traube C, Mauer EA, Gerber LM, Kaur S, Joyce C, Kerson A, Carlo C, Notterman D, Worgall S, Silver G, Greenwald BM. Cost Associated With Pediatric Delirium in the ICU. Crit Care Med. 2016 Dec;44(12):e1175-e1179. doi: 10.1097/CCM.0000000000002004. PMID 27518377
- [Background] Lei L, Li Y, Xu H, Zhang Q, Wu J, Zhao S, Zhang X, Xu M, Zhang S. Incidence, associated factors, and outcomes of delirium in critically ill children in china: a prospective cohort study. BMC Psychiatry. 2023 Dec 11;23(1):925. doi: 10.1186/s12888-023-05406-3. PMID 38082396
- [Background] Dervan LA, Di Gennaro JL, Farris RWD, Watson RS. Delirium in a Tertiary PICU: Risk Factors and Outcomes. Pediatr Crit Care Med. 2020 Jan;21(1):21-32. doi: 10.1097/PCC.0000000000002126. PMID 31568239
- [Background] Khan S, Haseeb A, Khalid M, Sher A, Haque A. Frequency and risk factors of delirium in the pediatric intensive care unit of a tertiary care hospital: A prospective observational study. Journal of pediatric critical care. 2024;11(1):10-4.